CLINICAL TRIAL: NCT00006309
Title: Pooling of Cohort Studies on Diet & Coronary Disease
Status: Completed | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Other Study IDs: 917; R01HL058904 (NIH)
Record Dates: First submitted 2000-09-28; First posted 2000-09-29 (Estimated); Last update posted 2016-02-18 (Estimated); Status verified 2004-12

CONDITIONS: Coronary Arteriosclerosis; Cardiovascular Diseases; Heart Diseases
MeSH Terms: conditions — Coronary Artery Disease; Cardiovascular Diseases; Heart Diseases

SUMMARY:
To quantify the role of dietary factors in the etiology of coronary heart disease by pooling data from 10 major prospective studies on diet and coronary heart disease.

DETAILED DESCRIPTION:
DESIGN NARRATIVE:

Specific hypotheses tested included an adverse effect of saturated fat and carotenoids (alpha-carotene, lutein, and lycopene), flavonoids, folic acid, and vitamin B6. Plausible biological interactions between nutrients, such as fatty acids of the n-6 and n-3 series were also explored. Each participating center sent data on tape to the coordinating unit at the Department of Nutrition, Harvard School of Public Health. The relations of dietary factors and coronary heart disease were first estimated within each study and compared for consistency. Data were then combined to obtain the best overall estimates, taking into account the validity of dietary data collected at each center. Members from study centers met annually to discuss the interpretation of findings. Over 6,000 cases of myocardial infarction or coronary death were anticipated, which should have provided excellent precision in measuring associations, and allowed the comparison of extreme intakes that were poorly represented in individual studies.

The study completion date listed in this record was obtained from the "End Date" entered in the Protocol Registration and Results System (PRS) record.

ELIGIBILITY:
No eligibility criteria

Max Age: 100 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 1999-09; Study Completion 2002-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alberto Ascherio — Harvard Medical School (HMS and HSDM)

REFERENCES:
- [Background] Pereira MA, O'Reilly E, Augustsson K, Fraser GE, Goldbourt U, Heitmann BL, Hallmans G, Knekt P, Liu S, Pietinen P, Spiegelman D, Stevens J, Virtamo J, Willett WC, Ascherio A. Dietary fiber and risk of coronary heart disease: a pooled analysis of cohort studies. Arch Intern Med. 2004 Feb 23;164(4):370-6. doi: 10.1001/archinte.164.4.370. PMID 14980987
- [Background] Knekt P, Ritz J, Pereira MA, O'Reilly EJ, Augustsson K, Fraser GE, Goldbourt U, Heitmann BL, Hallmans G, Liu S, Pietinen P, Spiegelman D, Stevens J, Virtamo J, Willett WC, Rimm EB, Ascherio A. Antioxidant vitamins and coronary heart disease risk: a pooled analysis of 9 cohorts. Am J Clin Nutr. 2004 Dec;80(6):1508-20. doi: 10.1093/ajcn/80.6.1508. PMID 15585762